CLINICAL TRIAL: NCT03085875
Title: POWERMOM, A Healthy Pregnancy Research Community
Status: Recruiting | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-17-6924
Record Dates: First submitted 2017-03-06; First posted 2017-03-21 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Pregnancy Related; Weight Change, Body; Health Problems in Pregnancy; Behavior
Keywords: Weight Change; Healthy Pregnancy; Physiologic Sensors
MeSH Terms: conditions — Body Weight Changes; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will take advantage of the open source framework of ResearchKit developed by Apple to bring research directly to participants. Using the ResearchKit platform as well as a stand alone app available for Android and HTML, it makes it easier to enroll large numbers of participants and carry out real-world health research to answer questions important to a broad population.

DETAILED DESCRIPTION:
* Eligibility determined, Individuals enrolled and consented to join study
* Short Intake Survey (demographic and baseline health information collected)
* Health History Survey (two days after participant enrolls in the study)
* Survey questions about current health and medical history will be sent to participants weekly. If participants had a prenatal visit during the week, a few additional questions will be asked.
* Twins / Multiples survey will begin appearing when a participant indicates they are having more than one baby
* Participants can submit home measurements of, weight and blood pressure as frequently as they want through HealthKit.
* Pregnancy outcome variables. (Miscarriage, stillbirth, birth of healthy baby, or pregnancy ended) will also be asked weekly.
* If the baby is born, questions about labor and delivery, as well as weight, size and birth date of the baby will be asked. A reminder to fill out the outcome survey will be given 4 weeks after a user's due date.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 16 years of age or older
* Pregnant women or within 8 weeks postpartum
* Currently live within the United States
* Own, and comfortable using, a smartphone or tablet

Exclusion Criteria:

• Inability to consent

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women, 16 years or older, who currently live in the United States, and own a smartphone.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2017-03-16 (Actual); Primary Completion 2027-03-13 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Improve our understanding of healthy pregnancy weight gain for all women. | Up to 46 weeks.
  Weight (lbs.) will be collected using surveys and measured with home and medical office scales.
Improve our understanding of how different factors impact pregnancy complications. | Up to 46 weeks.
  Pregnancy complications will be collected using surveys.
Improve our understanding how different factors impact the birth of the baby. | Up to 46 weeks.
  Birth outcomes will be collected using surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Lase Ajayi, MD, Principal Investigator — The Scripps Research Institute
Locations (1):
- Scripps Research Translational Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ajayi T, Kueper J, Ariniello L, Ho D, Delgado F, Beal M, Waalen J, Baca Motes K, Ramos E. Digital Health Platform for Maternal Health: Design, Recruitment Strategies, and Lessons Learned From the PowerMom Observational Cohort Study. JMIR Form Res. 2025 Apr 7;9:e70149. doi: 10.2196/70149. PMID 40194282
- See also: This study is being conducted online through the MyDataHelps app, study code PWRMOM — https://powermom.scripps.edu/